CLINICAL TRIAL: NCT05101811
Title: Assessment of Serum Vitamin D Levels in Women With Polycystic Ovary Syndrome
Brief Title: Vitamin D Levels in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ghamra Military Hospital (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Osama Mansour Khalifa Mohamed, Principal investigator,obstetrics and gynecologydepartment, Ghamra Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GhamraMH
Record Dates: First submitted 2021-10-08; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Control women without polycystic ovary syndrome (Experimental): Normal fertile women without polycystic ovary syndrome
  Interventions: Drug: Vitamin D Levels measurement using chemiluminescent assay; Device: Vitamin D level assessment
- Case women with polycystic ovary syndrome (Experimental): Women with polycystic ovary syndrome
  Interventions: Drug: Vitamin D Levels measurement using chemiluminescent assay; Device: Vitamin D level assessment

INTERVENTIONS:
Drug: Vitamin D Levels measurement using chemiluminescent assay — Measurement of serum vitamin D levels
Device: Vitamin D level assessment — Using lIAISON DEVICE

SUMMARY:
Polycystic ovary syndrome is the commonest endocrinopathy among women of reproductive age. Its worldwide prevalence has been estimated between5-10%.

Vitamin D, a fat-soluble vitamin, can be produced in two ways: by intestinal absorption and endogenous synthesis from a precursor of 17-hydroxyl cholesterol on the skin with sufficient exposure to ultraviolet sunlight.

DETAILED DESCRIPTION:
The aim of this work is assessment of the level of vitamin D in female have polycystic ovary syndrome & healthy female.and also make diagnostic criteria for patient who is in need for supplementations with vitamin D.

ELIGIBILITY:
Inclusion criteria:

* Hyperandrogenism
* Polycystic ovary syndrome

Exclusion Criteria:

* Thyroid disease
* Parathyroid disease
* Diabetes Mellitus
* Cushing syndrome
* Congenital adrenal hyperplasia
* Hyperprolactinemia
* Renal, liver or chronic disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Levels of vitamin D in Polycystic ovary syndrome | 1 year
  vitamin D levels is assumed to be significantly decreased

SECONDARY OUTCOMES:
Levels of vitamin D in fertile women | 1 year
  vitamin D level is expected to be normal

CONTACTS AND LOCATIONS:
Overall Officials: Osama Mohamed, Principal Investigator — Ghamra Military Hospital
Locations (1):
- Misr Al Gadida Military hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Summary and results
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year
Access Criteria: Al Azhar International Medical Journal
URL: https://aimj.journals.ekb.eg/